CLINICAL TRIAL: NCT01146119
Title: A Phase II, Randomized, Two Stage, Double-Blind, Placebo-Controlled, Safety and Immunogenicity Study of an Intramuscular Influenza Vaccine (Multimeric-001) Injected to Healthy Volunteers
Brief Title: Further Investigation of an Intramuscular Influenza Vaccine (Multimeric-001)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BiondVax Pharmaceuticals ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BVX-004
Record Dates: First submitted 2010-06-13; First posted 2010-06-17 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Influenza
Keywords: HAI; Influenza; prime; boost; immune response; seroconversion; universal; vaccine
MeSH Terms: conditions — Influenza, Human; HIV Seropositivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Multimeric-001, Adjuvanted (Experimental): 64 subjects received 2 injections of Adjuvanted Multimeric-001, 500 mcg with an interval of 21 days and then 60 days later were further immunized with a 15% dose of commercial seasonal trivalent vaccine (season 2011).
  Interventions: Biological: Multimeric-001, 500 mcg
- PBS and TIV 15% (Active Comparator): 32 subjects received 2 injections of PBS (Phosphate Buffered Saline) with an interval of 21 days and then were further immunized 60 days later with a 15% dose of commercial seasonal trivalent vaccine (season 2011).
  Interventions: Biological: PBS and TIV 15%
- Placebo, Adjuvanted (Placebo Comparator): 32 subjects received Adjuvanted PBS (Placebo) with an interval of 21 days.
  Interventions: Biological: Adjuvanted PBS
- Co-administration M-001 and TIV 15% (Experimental): 24 subjects received 2 injections on the same day, one injection containing Adjuvanted Multimeric-001 500 mcg and the other containing TIV 15%.
  Interventions: Biological: Multimeric-001, 500 mcg
- Co administration of M-001 and TIV 50% (Experimental): 24 subjects received 2 injections on the same day, one injection containing Adjuvanted Multimeric-001 500 mcg and the other containing TIV 50%.
  Interventions: Biological: Multimeric-001, 500 mcg
- Co administration of PBS and TIV 50% (Active Comparator): 24 subjects received 2 injections on the same day, one injection containing PBS and the other containing TIV 50%.
  Interventions: Biological: PBS and TIV 50%

INTERVENTIONS:
Biological: Multimeric-001, 500 mcg — Adjuvanted Multimeric-001 was administered twice with an interval of 19-23 days.
  Arms: Co administration of M-001 and TIV 50%; Co-administration M-001 and TIV 15%; Multimeric-001, Adjuvanted
Biological: Adjuvanted PBS — Adjuvanted PBS was administered twice with an interval of 19-23 days.
  Other Names: placebo
  Arms: Placebo, Adjuvanted
Biological: PBS and TIV 15% — PBS (Phosphate Buffered Saline) was administered twice with an interval of 19-23 days and then 60 days later a 15% dose of commercial seasonal trivalent vaccine (season 2011) was administered.
  Arms: PBS and TIV 15%
Biological: PBS and TIV 50% — PBS (Phosphate Buffered Saline) was administered twice with an interval of 19-23 days and then 60 days later a 50% dose of commercial seasonal trivalent vaccine (season 2011) was administered.
  Arms: Co administration of PBS and TIV 50%

SUMMARY:
This is a multi-center, randomized, two stage, double-blind, placebo-controlled administration study comprising 200 healthy participants.

DETAILED DESCRIPTION:
This is a Phase II multi-center, randomized, two stage, double-blind, placebo-controlled study comprising 200 participants. Eligible subjects will be randomized to receive one of the following administrations (as two single IM injections with an interval of 21 days between each injection Administration A: Prime twice with Adjuvanted Multimeric-001 500 mcg - 64 subjects.

Administration B: PBS (Placebo) twice - 32 subjects. Administration C: Adjuvanted PBS (Placebo)twice - 32 subjects. Participants from administrations A and B will be further immunized with a 15% dose of commercial seasonal trivalent vaccine for 2011 on day 81.

Administration D: Adjuvanted Multimeric-001 500 mcg coadministered once with 15% of TIV dose - 24 subjects. Administration E: Adjuvanted Multimeric-001 500 mcg coadministered once with 50% of TIV dose - 24 subjects Administration group F: PBS (Placebo) co-administered once with 50% of TIV dose - 24 subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females between the age of 18 and 49 years (inclusive).
* Subjects who provide written informed consent to participate in the study.
* Subjects able to adhere to the visit schedule and protocol requirements and be available to complete the study.
* Haematology, chemistry and urinalysis values with no clinical significance or do not reflect a medical condition which, according to the physician's judgment, might confound the results of the study or pose additional risk to the subject by participation in the study.
* Female of childbearing age must agree to use an acceptable method of contraception and male subjects should use a condom throughout the study period (until termination visit) if female partner is not using an effective contraceptive method.
* Subjects who are seronegative to at least one of the strains included in the seasonal vaccine against influenza for 2011.

Exclusion Criteria:

* Known history of significant medical disorder, which in the investigator's judgment, might confound the results of the study or pose additional risk to the subject by participation in the study.
* Subjects with known Guillain Barré Syndrome in the past.
* Two or more hospitalizations within the last year prior to screening visit.
* Known bleeding disorders including hemophilia or thrombocytopenia, or treatment with anticoagulant therapy (risk of bleeding with intramuscular injection).
* Immunocompromised patients and those receiving concomitant immunosuppressive therapy; or other immune modulating drugs including chronic steroid treatment.
* Subjects who have been immunized with anti-influenza vaccine or infected by influenza virus within eight months prior to the screening visit.
* Administration of any vaccine 30 days before the screening visit.
* Known hypersensitivity to previous influenza vaccination.
* Use of an influenza antiviral medication within 4 weeks of vaccination.
* Known hypersensitivity and/or allergy to any drug or vaccine.
* Known hypersensitivity to egg proteins (eggs or egg products), chicken proteins, or any of the vaccine components.
* Known history of drug or alcohol abuse.
* Any clinically significant abnormality upon physical examination or in the clinical laboratory tests at screening visit which, according to the physician's judgment, might confound the results of the study or pose additional risk to the subject by participation in the study.
* Increased liver enzymes more than 2.5 times above the upper reference level.
* Positive serology for HIV, HCV antibody or HBsAg.
* Any acute medical situation (e.g. acute infection, ongoing flu symptoms) with or without fever within 48 hours of vaccination, which is considered of significance by the Principal Investigator.
* Pregnant or lactating women at entry to study and those who are unwilling to agree to continue to use acceptable methods of contraception for two months after completion of the study (if applicable).
* Positive blood pregnancy test on screening.
* Subjects who participated in any clinical study within 30 days prior to study entry
* Subjects who are non-cooperative or unwilling to sign consent form.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2010-07; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | From day 0 until day 221
  Number of Participants with Adverse Events possible/probably related to the study drug in each group were similar in the experimental and control groups.
Anti Multimeric-001 antibodies | 21 days after second immunization with M-001
  Direct Elisa assay to test the titer of human antibodies that recognize the Multimeric-001 protein. Humoral immunity was manifested 21 and 60 days post immunization by significantly elevated anti-M-001 IgG levels among subjects administered twice with adjuvanted M-001

SECONDARY OUTCOMES:
Hemagglutination Inhibition (HAI) test for anti influenza antibodies | 21 days post co administration of M-001 and TIV 50%
  The serum is tested for its ability to adhere to influenza virus and thus inhibit the Hemagglutination reaction. Adjuvanted M-001 co-administered with partial dose of TIV (Vaxigrip, 50%) was effective in enhancing immunity to influenza-related antigens, as manifested by increased HAI antibody responses toward viruses contained in the TIV as well as toward non-TIV virus strains.

OTHER OUTCOMES:
Cellular Immunogenicity | 21 days after co administration of M-001 and TIV 50%
  Elevated proliferation of lymphocytes following in vitro incubation with M-001. The proliferation was associated with IFN gamma secretion

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Atsmon, MD, Principal Investigator — Clinical Research Center, Tel-Aviv Sourasky Medical Center; Yosef Caraco, Phd, Principal Investigator — Clinical Research Center, Hadassah Medical Center, Jerusalem
Locations (2):
- Israel (2):
  - Clinical Research Center, Hadassah Medical Center, Jerusalem
  - Clinical Research Center, Tel-Aviv Sourasky Medical Center, Tel Aviv